CLINICAL TRIAL: NCT02849886
Title: Use of Genetically Modified T-lymphocytes Expressing the Inducible Human Caspase 9 Gene (iCASP9) and the Selection Gene ΔCD19 in Allogeneic Haematopoietic Transplantation.
Brief Title: T Lymphocytes (LT) Expressing iCASP9 and ΔCD19 in Allogeneic Haematopoietic Transplantation.
Acronym: Side_by_Cide
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: not enough recruitment because of new therapeutic alternatives
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Etablissement Français du Sang (Other); Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: N/2000/39-B
Record Dates: First submitted 2016-05-19; First posted 2016-07-29 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Graft Versus Host Disease; Hematological Malignancies
Keywords: GvHD; Suicide gene; Dimerizer drug AP1903; Hematological stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LT icasp9 ΔCD19 (cohort1) (Experimental): Injection T lymphocytes iCASP9 ΔCD19 (2.10e6, 5.10e6 and 10.10e6 Gene Modified Cells (GMC)/kg).
  Interventions: Drug: T lymphocytes iCASP9 ΔCD19
- LT iCASP9 ΔCD19 & GvHD (cohort2) (Experimental): Injection T lymphocytes iCASP9 ΔCD19 (2.10e6, 5.10e6 and 10.10e6 GMC/kg). Patients who develop GVHD after administration of Gene Modified Cells (GMC) will be treated with dimerizer drug (AP1903)
  Interventions: Drug: T lymphocytes iCASP9 ΔCD19; Drug: Dimerizer drug AP1903

INTERVENTIONS:
Drug: T lymphocytes iCASP9 ΔCD19 — Intravenous injection of the T lymphocytes armed with the iCASP9 suicide gene
  Other Names: T lymphocytes Gene Modified Cells (GMC)
Drug: Dimerizer drug AP1903 — AP1903 drug will be administrated at a dose of 0.4 mg/kg by intravenous route in the two following cases:
  * Acute Grade ≥II or symptomatic Grade I GvHD justifying systemic immunosuppression therapy;
  * Grade ≥3 toxicity attributable to GMC.
  Other Names: Dimerizer drug
  Arms: LT iCASP9 ΔCD19 & GvHD (cohort2)

SUMMARY:
This study evaluates the frequency of occurrence, severity, and response to treatment by a chemical agent, notably the dimerizer AP1903 (Bellicum Pharmaceuticals compagny), in the case of acute Graft versus Host Disease (aGvHD) occurring after the administration of T-lymphocytes expressing iCASP9 and concomitantly to a bone marrow graft depleted in B- and T-lymphocytes

DETAILED DESCRIPTION:
Haematopoietic transplantation may result in serious complications, notably graft versus host disease (GvHD).

T-lymphocyte depletion of the bone marrow graft is able to prevent GvHD, while increasing the risk of rejection and reducing the antileukaemic effect of the graft (graft versus leukaemia, GvL). In a previous study, the investigators showed that the ex vivo transfer of the Herpes simplex thymidine kinase suicide gene (HSV-TK) into the graft's T lymphocytes prior to reinjection was not associated with immediate toxicity, while allowing for the prolonged recirculation of genetically modified cells (GMC) and control of induced GvHD by ganciclovir (GCV). In addition, this study revealed the existence of GMC resistant to GCV, an immunodeficiency of transduced cells, as well as an increased risk of Epstein-Barr virus (EBV)-induced lymphoproliferative disease. To overcome these difficulties, investigators improved the methodology of producing GMC by using a new vector (pMSCV-iCASP9-2A-ΔCD19) whose susceptibility gene was of human origin and associated with a human surface marker (non-functional) enabling the cell selection process. Moreover, the demonstration that the induced GvHD in this setting could be controlled by the administration of GCV alone led to significantly increase the number of genetically modified T-lymphocytes administered and omit cyclosporin prophylaxis of GvHD.

This phase I study will include 12 patients and will be conducted according the dose escalation method (2.10e6, 5.10e6 and 10.10e6 GMC / kg respectively for levels I, II & III). GMC will be prepared in the Cell and Tissue Engineering Laboratory (advanced therapy medicinal products departement) of the french Blood center (EFS) in Besançon, France, and sent to the transplantation department.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≤55 years (40< age ≤55 years);
* Patients who are candidates for myeloablative allogeneic bone marrow transplants: de novo or secondary acute lymphoblastic leukaemia (ALL) and acute myeloblastic leukaemia (AML) in complete remission (CR) ≥1; chronic myeloid leukaemia (CML) in chronic phase or in escape from tyrosine kinase inhibitors; myelodysplastic syndrome (MDS) with int-2 or high International Prognostic Scoring System (IPSS score, with medullary blastosis >10%); chemosensitive malignant non-Hodgkin's lymphoma (MNHL) in CR or partial remission (PR) >2 ; chemosensitive Hodgkin's disease in CR or PR >2 ; chemosensitive chronic lymphoid leukaemia (CLL) in CR or PR >2; chemosensitive myeloma in CR or PR ≥2;
* At high risk for GvHD: the risk for GvHD is considered high and the patient thus eligible for the study, if the receiver is >40 years, or if the donor is a woman and the receiver a man, regardless their age;
* Karnofsky index >70% or World Health Organization (WHO) index ≥2;
* Stable clinical conditions and life expectancy >3 months;
* Absence of organic disease contraindicating the transplantation
* Availability of a genotypically identical donor, aged >18 years, having given consent, and presenting no contraindications to bone marrow donation under general anaesthesia and to the required apheresis procedures;
* Written informed consent of the donor and patient.

Exclusion Criteria:

* Age <40 years or > 55 years
* Organic disease contraindicating the utilisation of myeloablative conditioning
* History of allogeneic Hematological Stem Cell Transplantation (HSCT);
* History of autologous HSCT <1 year prior to the date for the scheduled allogeneic HSCT;
* Neurological location of the haemopathy justifying the transplantation;
* Pregnant or breastfeeding woman;
* Positive HIV serology;
* Positive hepatitis B or hepatitis C serology (except for post-vaccinal hepatitis B status);
* Absence of informed consent from the receiver or donor;
* Inability to adhere to the protocol instructions.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-12-26 (Actual); Study Completion 2021-12-26 (Actual)

PRIMARY OUTCOMES:
GvHD response to Dimerizer AP1903 | 72 hours after administration of Dimerizer AP1903
  Disappearance of clinical signs of GvHD

SECONDARY OUTCOMES:
Haematopoietic reconstitution (Blood) | 1 month, 3 months, 6 months, and 1 year
  Full Blood count and Blood Cell phenotyping (T & B Lymphocytes, Natural Killers cells (NK), polynuclear cells...)
  Hematopoietic reconstitution will be assessed when % of Blood cells reach normal account values.
Haematopoietic engraftment (bone marrow) | 1 month, 3 months, 6 months, and 1 year
  Bone marrow smear analysis.
  Haematopoietic engraftment will be assessed when proportion of marrow cells reach normal account values.
Haematopoietic engraftment (chimerism) | 1 month, 3 months, 6 months, and 1 year
  Chimerism Analysis by quantitative mesurement (mesure of % of Donor & recipient cells)
  Full chimerism will be assessed when chimerim will reach 100% of donor profile.
Infections post Transplantation | 1 month, 3 months, 6 months, and 1 year
  Monitoring of Infections post-transplantation will be studied by analysis of frequency of infection's events.
  (number of infection's events by patients and/or frequency)
GvL effect | 1 month, 3 months, 6 months, and 1 year
  Molecular residual disease (MRD) analysis of biological markers of the initial hematological disease either by molecular biology and/or flow cytometry.
  GvL effect will be assessed by evaluation of decrease of initial tumoral load.

CONTACTS AND LOCATIONS:
Overall Officials: DECONINCK Eric, MD, PhD, HDR, Principal Investigator — CHRU de Besançon; Christophe FERRAND, PhD, HDR, Study Chair — EFSBFC-INSERM UMR1098; Marina DESCHAMPS, PhD, Study Chair — EFSBFC-INSERM UMR1098
Locations (1):
- CHU Jean Minjoz, Besançon, France

IPD SHARING:
Plan to Share IPD: Yes